CLINICAL TRIAL: NCT06072768
Title: Using SMART Design to Develop Dynamic Treatment Regimens for Glucocorticoid Tapering
Brief Title: Dynamic Treatment Regiments for Glucocorticoid Tapering
Acronym: SMART-RA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: IMMA-010-21S; CX002430 (Other Grant/Funding Number: VA CSR&D)
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Disease-modifying anti-rheumatic drug; Oral prednisone; Dose reduction; Tapering
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Participants will be allocated to the 15-day strategy preferentially until enrollment goals have been met; once completing the 15-day strategy, many participants will also be eligible to complete the 150-day strategy, and may subsequently enroll in it if they wish.
Masking Description: None (open label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 15-day taper prednisone (Experimental): This will be for 30 days. Participants will be allocated to the 15-day strategy preferentially until enrollment goals have been met; once completing the 15-day strategy, many participants will also be eligible to complete the 150-day strategy, and may subsequently enroll in it if they wish. Participants that are not eligible for the 15-day strategy, but are eligible for the 150-day strategy, will be enrolled in the 150-day strategy.
  Interventions: Drug: 15-day taper prednisone
- 150-day taper prednisone (Experimental): This will be for 180 days. Participants who are not eligible for the 15-day strategy, but are eligible for the 150-day strategy, will be enrolled in the 150-day strategy.
  Interventions: Drug: 150-day taper prednisone

INTERVENTIONS:
Drug: 15-day taper prednisone — The 15-day taper group will assess the effect of an approximately 50% oral prednisone dose reduction over 15 days, and will be followed for an additional 15 days after the last dose reduction.
  Arms: 15-day taper prednisone
Drug: 150-day taper prednisone — The 150-day taper group will assess the effect of reducing oral prednisone by 1 milligram (mg) every 30 days over 150 days, and will be followed for an additional 30 days after the last dose reduction.
  Arms: 150-day taper prednisone

SUMMARY:
The purpose of this clinical trial is to better understand how people with rheumatoid arthritis (RA) respond to gradual dose reduction, or "tapering", of steroid medications like prednisone. Some people with RA have symptoms when steroid dose is reduced, while others don't. This trial will look at different patient characteristics, including levels of inflammation in the body, differences in the way the brain processes sensory information, and certain hormone levels, to help researchers better understand why different people have these different responses to steroid tapering.

The hypotheses include:

* Greater or equal to ( ) 30% of participants in each arm will develop taper intolerance (either subjective, objective, or both) during the study period
* Greater or equal to 60% of participants will reduce Glucocorticoid dose by at least 5 Milligrams per day during the study period

DETAILED DESCRIPTION:
This trial was changed, so that participants could participate remotely without coming into the clinic. For participants coming into the clinic, the clinical disease activity index (CDAI) will be used to measure objective intolerance to tapering.

For remote participants, the Rheumatoid Arthritis Disease Activity Index (RADAI) will be used instead of the CDAI.

ELIGIBILITY:
Inclusion Criteria:

Ability to read and speak English to allow for written informed consent and patient-reported outcomes measures.

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Ability to take oral medication and be willing to adhere to the study intervention regimen
* Diagnosis of rheumatoid arthritis by a medical provider, confirmed by checking medical records.
* Current use of an RA treatment regimen of both oral prednisone and 1 other Food and Drug Administration-approved disease-modifying antirheumatic drug (DMARD), with no change in this therapy over the past 90 days

  1. Eligible DMARDs include the following: hydroxychloroquine, sulfasalazine, methotrexate, leflunomide, etanercept, adalimumab, infliximab, golimumab, certolizumab pegol, abatacept, tocilizumab, sarilumab, rituximab, tofacitinib, baricitinib, upadacitinib
  2. Patients enrolling in the 15-day taper must be taking 7.5mg/day oral prednisone
  3. Patients enrolling in the 150-day taper must be taking 5mg/day oral prednisone

Exclusion Criteria:

Current or recent (past year) use of systemic glucocorticoid (oral, intravenous, or intramuscular administration) >2 weeks for an indication other than RA, to reduce risk of adverse health outcomes related to worsening of the indicated condition

* Patients with greater than moderate RA activity as determined by the Clinical Disease Activity Index or by rheumatologist assessment, given high likelihood of taper failure in this population due to increased RA activity alone.
* Pre-existing primary or secondary adrenal insufficiency diagnosed by a physician, given high risk of worsening with prednisone taper
* Treatment with another investigational drug or intervention within 90 days
* Pregnancy
* Self-reported medical or psychiatric conditions that in the judgment of study personnel would preclude participation in this study (e.g., schizophrenia, malignancy, psychosis, suicidal ideation, history of substance abuse; note that stable anxiety and depression are NOT exclusions)
* Current, recent (within the last 6 months), or habitual use of artificial nails or nail enhancements. (Artificial nails can influence pressure pain sensitivity at the thumbnail);
* Any impairment, activity, behavior, or situation that in the judgment of the study team would prevent satisfactory completion of the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with subjective taper intolerance | Day 30 (15-day taper) or day 180 (150-day taper group)
  Subjective intolerance, the first point when a participant replies elects to stop glucocorticoid taper due to associated symptoms. This will be assessed using a one-question questionnaire with binary "yes" and "no" responses.
Number of participants with objective taper intolerance | Day 30 (15-day taper) or day 180 (150-day taper group)
  The first point when a participant develops any one of: increased RA activity (either clinical disease activity index [CDAI] increase of >2, or rheumatoid arthritis disease activity index [RADAI] of 1.5); RA flare (either CDAI increase of >1, or RADAI increase of >1 at a time when participant classifies as flaring; Clinical adrenal insufficiency.
Net glucocorticoid dose reduction | Day 30 (15-day taper) or day 180 (150-day taper group)
  The difference (in mg/day) between a participant's prednisone dose at enrollment, and either (1) the dose at which participants first develop taper intolerance, or (2) the dose at the end of study involvement, if participants do not develop taper intolerance.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Wallace, MD MSc, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (2):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No